CLINICAL TRIAL: NCT04303000
Title: Increasing Naloxone Access for Persons Who Use Opioids: An Online Recruitment and Training Approach to Opioid Overdose Education and Naloxone Distribution
Brief Title: Increasing Naloxone Access for Persons Who Use Opioids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michelle Sisson, M.A., Doctoral Student, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-300004762
Record Dates: First submitted 2020-03-03; First posted 2020-03-10 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Naloxone
Keywords: Opioid overdose; Naloxone distribution; Narcan; Online training
MeSH Terms: conditions — Opiate Overdose | interventions — Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opioid Overdose Education and Naloxone Distribution (Experimental): Participants will engage in online audiovisual training focused on recognizing the signs of an opioid overdose and the procedural steps for how to administer naloxone. Participants randomized to this arm will be provided with a naloxone nasal spray kit (4mg).
  Interventions: Drug: Opioid Overdose Education with Naloxone Distribution
- Opioid Overdose Education (Active Comparator): Participants will engage in online audiovisual training focused on recognizing the signs of an opioid overdose and the procedural steps for how to administer naloxone. Participants randomized to this arm will receive information about pharmacies in their area where they can purchase a naloxone kit.
  Interventions: Drug: Opioid Overdose Education

INTERVENTIONS:
Drug: Opioid Overdose Education with Naloxone Distribution — Online audiovisual training focused on recognizing the signs of an opioid overdose and administering naloxone. Participants are provided with a naloxone kit.
  Other Names: Narcan
  Arms: Opioid Overdose Education and Naloxone Distribution
Drug: Opioid Overdose Education — Online audiovisual training focused on recognizing the signs of an opioid overdose and administering naloxone. Participants are provided with information on where they can obtain a naloxone kit.
  Other Names: Narcan
  Arms: Opioid Overdose Education

SUMMARY:
Deaths relating to opioid overdose have rapidly increased over the past two decades. Due to the serious public health concern of the opioid epidemic, federal agencies recommend employing various harm reduction interventions. The implementation of Opioid Overdose Education and Naloxone Distribution (OEND) programs is effective in reducing opioid overdose mortality, yet these programs do not reach many high-risk individuals. Traditionally, OEND program venues are found in large, urban medical centers, drug treatment facilities, and needle exchange programs. Identifying unreached, high-risk individuals and providing training and naloxone kits through online recruitment could significantly expand access to this life-saving intervention. The primary goal of the current proposed project is to examine the acceptability and feasibility of online recruitment, online opioid overdose and naloxone administration education, and postal distribution of naloxone kits.

DETAILED DESCRIPTION:
Drug overdose is the leading cause of accidental death in the United States, with over 65% of drug related fatalities resulting from the use of opioids. The continually increasing rates of opioid overdose deaths in the last two decades have led to the declaration of an opioid epidemic. Over a brief 15-year period, from 1999-2014, drug overdose related deaths tripled and rates have continued to sharply escalate since then. Federal agencies have responded to this crisis with various recommendations including enhancing harm reduction approaches such as naloxone distribution. Naloxone is an opioid antagonist that can be used to reverse opioid overdose. Though it is typically administered in Emergency Departments, laypersons have recently been successfully trained through Opioid Overdose Education and Naloxone Distribution (OEND) programs to recognize signs of opioid overdose and perform timely administration of naloxone in homes and community settings while awaiting medical services. Several studies have demonstrated that OEND programs effectively reduce opioid overdose mortality and are safe and cost-effective. However, OEND programs are typically implemented in urban areas as part of large medical center research programs, needle exchanges, or drug treatment programs. Individuals living in areas without these programs or services lack access to critical and life-saving OEND. The current proposal will examine the acceptability and feasibility of online recruitment, online opioid overdose education, and postal distribution of naloxone kits (N=80). Opioid users at risk for overdose will be recruited online through Craigslist. If eligible, participants will complete an opioid use questionnaire and will indicate if they are interested in receiving opioid overdose and naloxone administration training. If interested, they will complete pre- and post-intervention knowledge questionnaires, engage in audiovisual training, and half will be randomized to receive a naloxone kit in the mail while the other half will be given information on where they can receive a naloxone kit. All participants will complete remote follow-up assessments at 1, 2, and 3 months post study to evaluate naloxone kit use and outcomes. This study will evaluate a novel approach to providing OEND to individuals with otherwise limited access to this type of intervention. Successful implementation of remote OEND through this project would support future employment of similar remote programs to expand this critical harm reduction strategy to high-risk individuals in areas lacking traditional OEND programs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Current or past six months illicit use of opioids
* Electronic device access for online survey completion
* Willing to provide email address to receive survey link and compensation
* Able to read and speak English
* Willing to provide their contact information and that of two friends/family members
* Permanent address for mailing of naloxone kit
* Does not currently have a naloxone kit in possession

Exclusion Criteria:

* Contraindication for naloxone (known severe allergic reaction)
* Cognitive impairment or unstable psychiatric condition that interferes with the informed consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-07-11 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Sisson, MA, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - Craigslist, Anniston, Alabama
  - Craigslist, Gadsden, Alabama
  - Craigslist, Mobile, Alabama
  - Craigslist, Montgomery, Alabama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sisson ML, Azuero A, Hawes E, Chichester KR, Carpenter MJ, Businelle MS, Shelton RC, Cropsey KL. Characterizing Individuals Who Elect and Decline Opioid Overdose Education and Naloxone Distribution to Tailor Programs and Expand Impact. J Addict Med. 2025 May-Jun 01;19(3):268-273. doi: 10.1097/ADM.0000000000001407. Epub 2024 Nov 8. PMID 39514898
- [Derived] Sisson ML, Azuero A, Chichester KR, Carpenter MJ, Businelle MS, Shelton RC, Cropsey KL. Preliminary effectiveness of online opioid overdose and naloxone administration training and impact of naloxone possession on opioid use. Drug Alcohol Depend. 2023 Aug 1;249:110815. doi: 10.1016/j.drugalcdep.2023.110815. Epub 2023 Jun 7. PMID 37336007
- [Derived] Sisson ML, Azuero A, Chichester KR, Carpenter MJ, Businelle MS, Shelton RC, Cropsey KL. Feasibility and acceptability of online opioid overdose education and naloxone distribution: Study protocol and preliminary results from a randomized pilot clinical trial. Contemp Clin Trials Commun. 2023 Apr 5;33:101131. doi: 10.1016/j.conctc.2023.101131. eCollection 2023 Jun. PMID 37091508

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via online social media platforms (e.g., Craigslist) between July and October 2021.
Pre-assignment Details: A total of 13 participants were not randomized to a group for the training portion of the study, as they did not complete the baseline assessment.
Groups:
- Screened Participants: Started and completed screening
- Opioid Overdose Education and Naloxone Distribution: Participants engaged in online audiovisual training focused on recognizing the signs of an opioid overdose and the procedural steps for how to administer naloxone. Participants randomized to this arm were provided with a naloxone nasal spray kit (4mg).
  Opioid Overdose Education with Naloxone Distribution: Online audiovisual training focused on recognizing the signs of an opioid overdose and administering naloxone. Participants were provided with a naloxone kit.
- Opioid Overdose Education: Participants engaged in online audiovisual training focused on recognizing the signs of an opioid overdose and the procedural steps for how to administer naloxone. Participants randomized to this arm received information about pharmacies in their area where they could purchase a naloxone kit.
  Opioid Overdose Education: Online audiovisual training focused on recognizing the signs of an opioid overdose and administering naloxone. Participants were provided with information on where they could obtain a naloxone kit.
Period: Opioid Use Questionnaire
Arm/Group | Screened Participants | Opioid Overdose Education and Naloxone Distribution | Opioid Overdose Education
Started | 319 | 0 (Participants were randomized to group after the first study period.) | 0 (Participants were randomized to group after the first study period.)
Completed | 304 | 0 (The total number of participants who completed this period of the study is 304. Participants were randomized to groups after this study period.) | 0 (The total number of participants who completed this period of the study is 304. Participants were randomized to groups after this study period.)
Not Completed | 15 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 0 | 0
Period: Training Portion
Arm/Group | Screened Participants | Opioid Overdose Education and Naloxone Distribution | Opioid Overdose Education
Started | 0 | 55 | 56
Month 1 Follow-Up | 0 | 48 | 50
Month 2 Follow-Up | 0 | 48 | 50
Month 3 Follow-Up | 0 | 47 | 48
Completed | 0 | 45 | 47
Not Completed | 0 | 10 | 9

BASELINE CHARACTERISTICS:
Population: Baseline characteristics described here are for the 111 participants enrolled in the training portion of the study who were randomized to either the "Opioid Overdose Education and Naloxone Distribution" or "Opioid Overdose Education" groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid Overdose Education and Naloxone Distribution | Opioid Overdose Education | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.44 (9.08) | 38.54 (10.54) | 37.93 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 20 | 22 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 53 | 54 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 46 | 45 | 91
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 56 | 111

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants That Completed the Training in 6 Months
Description: Feasibility of online opioid overdose education and remote naloxone distribution as indicated by recruitment of at least 80 total participants in 6 months. There was not a calculated measure, and this aspect of feasibility was based on ability to recruit a set number of participants in a predetermined amount of time.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Overdose Education and Naloxone Distribution | Opioid Overdose Education
Number analyzed (Participants) | 55 | 56
Participants
  Enrolled and Randomized | 55 | 56
  Lost to Follow-up | 10 | 9

2. Primary Outcome: Change in Participant Knowledge of Opioid Overdose Response Procedures
Description: Mean change in participant knowledge as indicated by difference in scores on pre- and post-training knowledge questionnaires on a scale of 1 to 9 where 9 indicates greater knowledge.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opioid Overdose Education and Naloxone Distribution | Opioid Overdose Education
Number analyzed (Participants) | 55 | 56
score on a scale | 1.48 (1.83) | 1.34 (1.51)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were not collected during the pre-randomization period.
Arm/Group | Opioid Overdose Education and Naloxone Distribution | Opioid Overdose Education
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT04303000/Prot_SAP_002.pdf